CLINICAL TRIAL: NCT04389372
Title: Feasibility and Effectiveness of Mindfulness Program by Smartphone for Patients with Chronic Migraine and Medication Overuse During Covid-19 Emergency
Brief Title: Effectiveness and Acceptability of MINDFULNESS by Smartphone, for Patients with Chronic Migraine and Medication Overuse
Acronym: ChroMig-Smart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chro-Mig-Smart
Record Dates: First submitted 2020-05-05; First posted 2020-05-15 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness by Smartphone (Experimental): mindfulness therapy by smart phone
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness by smartphone combined to video calls for clinical evaluation in patients with chronic migraine and medication overuse after withdrawal program

SUMMARY:
Chronic Migraine is a disabling condition that affects the 2% of migraine population. It is often associated with medication overuse that makes this condition very difficult to treat. The literature of the last decades confirm the efficacy of withdrawal for patients with medication overuse but it is also confirmed that patients have to be carefully followed in the last period after withdrawal to avoid relapses and to improve the clinical benefit of the therapeutic approach. It has been also reported how the clinical results can be improved when traditional therapies are combined with behavioral approaches in particular mindfulness, that help patient to become more conscious about their symptoms and able to manage pain without medication. Generally patients after withdrawal follow a specific prophylaxis for migraine, but also come weekly to the hospital for practicing mindfulness for 6 sessionsAs the emergency situation due to the Corona-virus pandemic phenomenon in Italy, patients will miss the possibility to come for the regular practice to the hospital: for this reason the investigator propose a small pilot study to enforce the use of technology for our patients so that they can continue to be followed in their therapeutic process. This preliminary study will be conducted on 25 patients that have been submitted to a withdrawal according to the standard procedure at our hospital and they will practice mindfulness daily by a standard session of 12 minutes on their smartphone recorded by the expert who generally manage their sessions at the hospital and also a weekly video-call to evaluate the clinical condition and to encourage to use strategies for pain management. This modality will allow the patients to continue their therapeutic process and to be followed regularly during the one year after withdrawal

DETAILED DESCRIPTION:
Background and significance Chronic Migraine is a disabling condition that affects the 2% of migraine population. It is often associated with medication overuse that makes this condition very difficult to treat. The literature of the last decades confirm the efficacy of withdrawal for patients with medication overuse. Also, patients need to be carefully followed after withdrawal to avoid relapses in overuse and to improve the clinical benefit. It has been also reported that the clinical results can be improved if traditional therapies are combined with behavioral approaches in particular mindfulness, that help patients to become more conscious about their symptoms and able to manage pain without medication.

This preliminary study will be performed because the emergency for Covid-19 with the restrictions imposed will not allow patients. The literature of the last decades promote the use of smart phone or telemedicine for clinical and therapeutic application with encouraging results. Twenty five patients that have been submitted to a withdrawal according to the standard procedure at our hospital will practice mindfulness daily by a standard session of 12 minutes on their smartphone recorded by the expert who generally manage their sessions at the hospital. Also a weekly video-call to evaluate the clinical condition and to encourage to use strategies for pain management will be scheduled.

This modality will allow the patients to continue their therapeutic process and to be followed regularly during the one year after withdrawal

ELIGIBILITY:
Inclusion Criteria:+

1. Years age >18 yrs
2. clinical diagnosis of Chronic Migraine with medication Overuse
3. withdrawal treatment at the Besta institute
4. written informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of Mindfullness by Smartphone | at 6 months and 12 months follow-up compared with baseline (Headache Daily Diary)
  Changes in migraine /days per month and medication intake/month (decrease of at least 50% in at least 50% of CM-MO patients)

SECONDARY OUTCOMES:
Change of Disability Score | 6months - 12months
  Changes in disability, impact Migraine Disability Assessment Score (MIDAS questionnaire) minimum score 0-maximum score 270 HIGHER SCORES worse outcome (they indicate more disability)
Change in Quality of life | 6months - 12 months
  Changes in Headache Impact Test (HIT-6) minimum score 36- maximum score 78 HIGHER SCORES worse outcome (they indicate more impact)

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Neurologia 3, Milan, Milano, Italy

REFERENCES:
- [Derived] Rizzoli PB, Grazzi L. Adaptation of the management of chronic migraine patients with medication overuse to the suspension of treatment protocols during the COVID-19 pandemic: Lessons from a tertiary headache center in Milan-6-month results. Headache. 2021 Jun;61(6):961-962. doi: 10.1111/head.14140. Epub 2021 Jun 21. No abstract available. PMID 34153116